CLINICAL TRIAL: NCT03959956
Title: Community Use of Digital Auscultation to Improve Diagnosis of Pediatric Pneumonia in Sylhet, Bangladesh
Brief Title: Improving Paediatric Pneumonia Diagnosis Using Digital Auscultation
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Projahnmo Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PR-19004
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Childhood Pneumonia
Keywords: Digital auscultation; Pneumonia; Lung sounds; IMCI; LMIC
MeSH Terms: conditions — Pneumonia; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Recording lung sound by a Smartscope — Lung sound will be recorded from four chest points by an electronic stethoscope called Smartscope which can also classify the recorded lung sound.

SUMMARY:
This study aims to evaluate an automated interpretation algorithm of recorded lung sound by a digital stethoscope, name the Smartscope, among rural Bangladeshi children receiving community care in order to improve the diagnosis of childhood pneumonia at first level facility in low- and middle-income countries. A mixed-methods study will be conducted for a period of twelve months in rural Sylhet, Bangladesh. A total of 12 community health workers (CHWs) and 12 community healthcare providers (CHCPs) will be recruited and trained for this study. CHWs will conduct household surveillance to identify children with cough and difficult breathing and refer to nearby community clinic (CC). The CHCPs will screen the children at the CCs as per protocol and enroll the suspected cases with couth or difficult breathing. A total of 1003 children will be enrolled in this study. Enrolled children will be assessed for signs and symptoms of pneumonia including oxygen saturation. The children will have their lung sounds recorded by the Smartscope at four sequential locations. A listening panel comprises by pediatricians will generate one summary patient classification of normal, crackle, wheeze, crackle and wheeze, or uninterpretable. The Respiratory detector automated algorithm will be applied to the lung recording to generate an interpretation. The study hypothesis is more than 50% of patients will have quality lung sound recordings and the agreement between the automated computerized analysis by Respiratory Detector and an expert listening panel will be high (kappa >0.5).

DETAILED DESCRIPTION:
Background Childhood pneumonia is the second leading cause of under-five death accounting for about 0.921 million children globally.1 About 120 million new episodes of childhood pneumonia occur each year worldwide.2 The estimated incidence is 0.015 episodes per child-year in developed and 0.22 episodes per child-year in developing countries in this age group.3 In Bangladesh, the annual incidence of pneumonia is 36 per 100 child-years.4 Expanding pneumonia treatment beyond higher level facility and into first level facility settings with lay community health workers (CHWs) is an emerging strategy that can address gaps in care access. World Health Organization (WHO) recommended healthcare providers to use practical, standardised case management guidelines for childhood pneumonia care.5,6 However, these guidelines do not include lung auscultation in their pneumonia definition for frontline healthcare workers6 because of its high inter-observer variability and subjectivity, regardless of healthcare providers training level.7-11 Digital auscultation by electronic stethoscopes may overcome these limitations.

An innovative, low-cost digital auscultation device was developed especially for children called Smartscope. The Smartscope improves lung signal strength by uniformly distributing highly sensitive electret microphone arrays across the stethoscope diaphragm so that the entire audible spectrum can be captured, a critical feature for identifying higher frequency pathologic lung sounds. It's rechargeable battery can power >20 hours of use, important in rural communities with inconsistent electricity. The device mitigates movement artifact and tubular resonance by using an ergonomic design to better secure the device on the child's chest. It also eliminates the rubber stethoscope tubing, a source of ambient noise and friction contamination. It includes an integrated external microphone that removes unwanted ambient noises. The Smartscope also permits onboard data storage with a microSD card and is equipped with automated analysis software.12 Smartscope has been successfully validated in the laboratory against the Littmann 3200 electronic stethoscope and has demonstrated comparable results. This Smartscope has the potential to be a highly specific respiratory diagnostic tool that is feasible for use by community-based healthcare workers in LMICs. This project proposes to evaluate the potential impact of digital auscultation at first level facilities in rural Bangladesh.

Objectives

1. To assess whether lung sounds recorded using Smartscope in children by Community Health Care Provider (CHCP) at CC meet pre-defined quality thresholds established by experts.
2. Determine the reliability and performance of the Smartscope Respiratory Detector automated analysis algorithm on lung sounds recorded by CHCP using the Smartscope, compared to reference interpretations by a paediatric listening panel.
3. Collect hypothesis-generating pilot data on the impact of digital auscultation on treatment decision-making by CHCPs, assuming lung recordings as the reference, as well as document equipment usability and durability during the project in order to understand whether additional device refinements are necessary.
4. Determine the acceptability of the Smartscope among CHCP and carers of children evaluated with the Smartscope.

Methods A mixed-methods study will be conducted in rural Sylhet district of Bangladesh. Bangladesh has established about 13,000 CCs, one each for ~6,000 people. CCs are staffed by a CHCP with at least 12th-grade education and 3 months of pre-service training including Integrated Management of Childhood Illness (IMCI) guidelines. Twelve CCs will be selected purposively in Zakiganj and Kanaighat sub-districts of Sylhet district. Additionally, a total of 12 CHWs will be recruited and trained for this study. Each CHW will cover approximately ~13,000 population with ~1,400 under-five children. CHWs will visit each child aged 0-59 months in her catchment area every other month. The CHW will evaluate the child for signs/symptoms of pneumonia and question the mother or carer about any history of these symptoms. All suspected pneumonia cases (history/observed cough or difficult breathing) will be referred or accompanied to CCs with a referral slip for further evaluation and treatment. A study physician will be recruited for providing training and supervision of CHCPs and CHWs in clinical assessment, measurement of oxygen saturation and recording lung sound by the Smartscope.

Screening: CHCPs in the CC will screen all under-five children as per protocol using a screening form. Approximately 7,200 children will be screened. If the child becomes eligible, the carer will be invited for consent to participate in the study.

Enrolment: If the carer gives consent, the child will be enrolled in the study. A total of 1003 children with history/observation of cough or difficult breathing (possible pneumonia) will be enrolled.

Lung auscultation: Lung sounds will be recorded using Smartscope. It is being used for its intended purpose only.

1. Sound collection: Enrolled children will have their lung sounds recorded at four sequential locations (two anterior and two posterior chest positions) for ~10 seconds/position. The recording procedure lasts approximately 60 seconds and captures 3-4 full breath cycles/position. Daily or alternate day Smartscope lung sounds will be uploaded to a server and securely stored. Later on, this lung sounds will be processed and used by the personnel involved in this study.
2. Sound processing: A novel sound-filtering algorithm will be applied to lung recordings to reduce ambient noise and optimize lung sound quality.
3. Listening panel: Three practicing pediatricians will form the panel. One will serve as the arbitrator and two as primary listeners. All panelists will be trained and standardized to the methodology developed and validated during PERCH. Panelists will generate one summary patient classification of normal, crackle, wheeze, crackle and wheeze, or uninterpretable. Two primary listeners will independently classify the recorded lung sounds, any discrepancies will be resolved through discussion, and if not resolved then the third listener will arbitrate.
4. Respiratory detector: The Respiratory Detector automated algorithm will be applied to the lung recordings to generate an interpretation.

Pulse oximetry: Pulse oximetry will also be performed using a Masimo® Rad5 oximeter to all eligible consented children. If any child's oxygen saturation found <90% will be referred to the sub-district health center or Sylhet Osmani Medical College Hospital.

Collecting socioeconomic and confounders data: CHW will collect socio-economic and other related confounders' data including immunization information, weight, mid-upper arm circumference and length/height from all enrolled cases at the household level within seven days of enrolment.

Focus group discussions: Four focus group discussions (FGDs) will be organized, two with carers (one with female and one with male) and one with CHCPs and one with CC management committee members and community leaders to share their opinions about the Smartscope. Each FGD will consist of 8-12 participants. A trained moderator will lead the discussion about perceptions of the Smartscope and the acceptability of Smartscope as a diagnostic for pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 60 months
* History or observation of cough or difficult breathing
* Provide written informed consent

Exclusion Criteria:

* If enrolled within the last 30 days in this study
* Severely ill children who need to be referred immediately
* Refusal to join the study

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be children aged less than 60 months who will visit the community clinics of Zakiganj and Kanaighat Subdistrict of Sylhet, Bangladesh and identified as suffering from cough or difficult breathing.
Sampling Method: Probability Sample
Enrollment: 990 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Quality of lung sound recording by healthcare worker | At the time of enrollment
  Quality lung sound recordings using pre-determined quality metrics i.e., at least 75% interpretable lung sound segments per patient (3 out of 4 chest positions). and high between listener agreement for the presence or absence of abnormal lung sounds (kappa>0.8).
Performance of the automated analysis of lung sound | within 3 months after collection of recorded lung sound
  It will be evaluated comparing with listener interpretation of classification of lung sound; assuming agreement will be high (kappa>0.6)

CONTACTS AND LOCATIONS:
Locations (1):
- Zakiganj Upazila Health Complex, Sylhet, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu L, Oza S, Hogan D, Chu Y, Perin J, Zhu J, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of under-5 mortality in 2000-15: an updated systematic analysis with implications for the Sustainable Development Goals. Lancet. 2016 Dec 17;388(10063):3027-3035. doi: 10.1016/S0140-6736(16)31593-8. Epub 2016 Nov 11. PMID 27839855
- [Background] Walker CLF, Rudan I, Liu L, Nair H, Theodoratou E, Bhutta ZA, O'Brien KL, Campbell H, Black RE. Global burden of childhood pneumonia and diarrhoea. Lancet. 2013 Apr 20;381(9875):1405-1416. doi: 10.1016/S0140-6736(13)60222-6. Epub 2013 Apr 12. PMID 23582727
- [Background] Rudan I, O'Brien KL, Nair H, Liu L, Theodoratou E, Qazi S, Luksic I, Fischer Walker CL, Black RE, Campbell H; Child Health Epidemiology Reference Group (CHERG). Epidemiology and etiology of childhood pneumonia in 2010: estimates of incidence, severe morbidity, mortality, underlying risk factors and causative pathogens for 192 countries. J Glob Health. 2013 Jun;3(1):010401. doi: 10.7189/jogh.03.010401. PMID 23826505
- [Background] Margolis PA, Ferkol TW, Marsocci S, Super DM, Keyes LL, McNutt R, Harrell FE Jr. Accuracy of the clinical examination in detecting hypoxemia in infants with respiratory illness. J Pediatr. 1994 Apr;124(4):552-60. doi: 10.1016/s0022-3476(05)83133-6. PMID 8151469
- [Background] Murphy RL, Vyshedskiy A, Power-Charnitsky VA, Bana DS, Marinelli PM, Wong-Tse A, Paciej R. Automated lung sound analysis in patients with pneumonia. Respir Care. 2004 Dec;49(12):1490-7. PMID 15571639
- [Background] Grenier MC, Gagnon K, Genest J Jr, Durand J, Durand LG. Clinical comparison of acoustic and electronic stethoscopes and design of a new electronic stethoscope. Am J Cardiol. 1998 Mar 1;81(5):653-6. doi: 10.1016/s0002-9149(97)00977-6. PMID 9514471
- [Background] Brooks D, Thomas J. Interrater reliability of auscultation of breath sounds among physical therapists. Phys Ther. 1995 Dec;75(12):1082-8. doi: 10.1093/ptj/75.12.1082. PMID 7501711
- [Background] Gjlrup T, Bugge PM, Jensen AM. Interobserver variation in assessment of respiratory signs. Physicians' guesses as to interobserver variation. Acta Med Scand. 1984;216(1):61-6. doi: 10.1111/j.0954-6820.1984.tb03772.x. PMID 6485882
- [Background] Emmanouilidou D, McCollum ED, Park DE, Elhilali M. Computerized Lung Sound Screening for Pediatric Auscultation in Noisy Field Environments. IEEE Trans Biomed Eng. 2018 Jul;65(7):1564-1574. doi: 10.1109/TBME.2017.2717280. Epub 2017 Jun 19. PMID 28641244
- [Derived] Ahmed S, Mitra DK, Nair H, Cunningham S, Khan AM, Islam AA, McLane IM, Chowdhury NH, Begum N, Shahidullah M, Islam MS, Norrie J, Campbell H, Sheikh A, Baqui AH, McCollum ED. Digital auscultation as a novel childhood pneumonia diagnostic tool for community clinics in Sylhet, Bangladesh: protocol for a cross-sectional study. BMJ Open. 2022 Feb 9;12(2):e059630. doi: 10.1136/bmjopen-2021-059630. PMID 35140164